CLINICAL TRIAL: NCT05585749
Title: The Effect of Virtual Reality Application on Pain Intensity and Anxiety Level in Endoscopy Patients
Brief Title: Virtual Reality Application on Pain Intensity and Anxiety Level in Endoscopy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/ 04 - 22
Record Dates: First submitted 2022-09-22; First posted 2022-10-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: Virtual Reality; Anxiety; Pain; Endoscopy Patients
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Virtual Reality Based Relaxation Program
Who Masked: Participant
Masking Description: Virtual Reality Based Relaxation Program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Based Relaxation Program (Experimental): Virtual Reality Based Relaxation Program
  Interventions: Other: Virtual Reality Based Relaxation Program
- Control group (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Other: Virtual Reality Based Relaxation Program — Virtual Reality Based Relaxation Program
  Arms: Virtual Reality Based Relaxation Program

SUMMARY:
In contemporary medicine, endoscopic procedures are often regarded as the gold standard for the diagnosis and treatment of gastrointestinal illnesses due to the essential role they play in these processes. Endoscopy is a minimally invasive procedure that allows direct visualization of the gastrointestinal tract using a flexible, camera-equipped instrument.However, due to their invasive nature, these methods pose certain challenges for both healthcare professionals and patients. In particular, the physical discomfort and pain experienced during the procedure can lead to a negative attitude toward the process in patients, which can indirectly affect the success of the procedure .Despite the fact that a number of studies have examined the impact of virtual reality applications on pain and anxiety during endoscopy, the conclusions remain inconsistent. Moreover, relatively few studies have assessed physiological signs of anxiety. Therefore, uncertainties remain regarding the generalizability of existing findings. The present study aimed to examine the effect of virtual reality application on pain, anxiety, and physiological parameters in patients undergoing endoscopy.

ELIGIBILITY:
Eligible individuals were adults aged 18 or older, capable of effective communication, and scheduled for non-sedated oral gastroduodenoscopy (OGD).

Exclusion criteria included emergency endoscopy, neurological conditions (e.g., migraine, vertigo, chronic headaches), or sensory impairments affecting hearing or vision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 hours later
  Visual Analog Scale is used to convert some values that cannot be measured numerically into digital. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing.0 points means no pain, 100 points means a lot of pain
Anxiety Assessment Scale | 1 hours later
  Patients will be asked to show their anxiety levels before and after the procedure on a 10 cm long horizontal line. Line has 0 at the beginning and 10 at the end. 10 means very extreme anxiety and 0 means no anxiety.
Physiological Symptoms of Anxiety Follow-up Form | 1 hours later
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation value.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bahçecioğlu Turan, PhD, Study Chair — Firat University
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No